CLINICAL TRIAL: NCT02457650
Title: Phase I Study of Malignancies That Express NY-ESO-1 With T Cell Receptor-transduced T Cells Targeting NY-ESO-1
Brief Title: T Cell Receptor-transduced T Cells Targeting NY-ESO-1 for Treatment of Patients With NY-ESO-1- Expressing Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: Shenzhen Institute for Innovation and Translational Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504002
Record Dates: First submitted 2015-05-12; First posted 2015-05-29 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Bladder Carcinoma; Breast Cancer; Esophagus Carcinoma; Lung Cancer; Melanoma; Multiple Myeloma; Neuroblastoma; Ovarian Cancer; Synovial Sarcoma; Other Metastatic Solid Cancers
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Esophageal Neoplasms; Lung Neoplasms; Melanoma; Multiple Myeloma; Neuroblastoma; Ovarian Neoplasms; Sarcoma, Synovial | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-NY ESO-1 TCR-transduced T cells (Experimental): Patients will receive a lymphodepleting conditioning regimen followed by an infusion of anti-NY-ESO-1 TCR-transduced T cells.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Anti-NY ESO-1 TCR-transduced T cells

INTERVENTIONS:
Drug: Cyclophosphamide — On days -7 through -6, Cyclophosphamide 60mg/kg/day IV will be infused over 60 minutes.
Drug: Fludarabine — On days -5 through -1, Fludarabine 25mg/m2/day IV will be infused over 30 minutes.
Biological: Anti-NY ESO-1 TCR-transduced T cells — Modified cells will be infused IV over 30 minutes.

SUMMARY:
Background:

Autologous T cells engineered to express a T cell receptor (TCR) targeting NY-ESO-1 will be infused back to patients with NY-ESO-1- expressing malignancies. The patients pretreated with a lymphodepleting preconditioning regimen will be monitored after infusion of anti-NY-ESO-1 TCR-transduced T cells for adverse events, persistence of anti-NY-ESO-1 TCR-transduced T cells and treatment efficacy.

Objectives:

To evaluate the safety and the efficacy of anti-NY-ESO-1 TCR-transduced T cell-based immunotherapy for patients with NY-ESO-1- expressing malignancies.

Eligibility:

Patients older than one year of age, who have relapsed or refractory malignancies that express both NY-ESO-1 and human leukocyte antigen (HLA)-A2 molecules.

Patients must have adequate organ functions.

Design:

* Peripheral blood from patients will be collected for isolation of peripheral blood mononuclear cells (PBMCs), which will be transduced with a lentiviral or retroviral vector encoding an HLA-A2 restricted anti-NY-ESO-1 TCR gene.
* Patients will receive a lymphodepleting preconditioning regimen to prepare their immune system to accept modified T cells.
* Patients will receive an infusion of their own modified T cells. They will remain in the hospital to be monitored for adverse events until they have recovered from the treatment.
* Patients will have frequent follow-up visits to monitor the persistence of modified T cells and efficacy of the treatment.

DETAILED DESCRIPTION:
Despite advances has been made to date in the treatment of patients with hematologic malignancies, clinical trials targeting solid cancers have achieved limited efficacy. One important reason is due to lack of ideal cancer antigens. NY-ESO-1 is expressed in various types of cancers, including neuroblastoma, hepatoma, myeloma, melanoma, esophagus, prostate, bladder, breast and ovarian cancers. While, in normal somatic tissues, NY-ESO-1 expression is restricted to the germline cells, which lack HLA molecules and cannot present peptides derived from NY-ESO-1 for recognition by T cells. Therefore, NY-ESO-1 specific T cells will only recognize and kill NY-ESO-1-expressing cancer cells, but not normal cells, thus avoiding induction of autoimmune reaction. With these unique features, NY-ESO-1 has been selected as an attractive tumor antigen candidate for cancer immunotherapy in various clinical trials.

In this trial, autologous T cells engineered to express a T cell receptor (TCR) targeting NY-ESO-1 will be infused back to patients with NY-ESO-1- expressing malignancies after they receive a lymphodepleting preconditioning regimen. The patients will be monitored after infusion of anti-NY-ESO-1 TCR-transduced T cells for adverse events, persistence of anti-NY-ESO-1 TCR-transduced T cells and treatment efficacy.

Primary objectives:

To determine the safety and feasibility of the administration of anti-NY-ESO-1 TCR transduced T cells in patients with HLA-A2+ NY-ESO-1-expressing malignancies.

Secondary objectives:

To determine if the treatment can result in clinical regression of malignant tumors in the patients.

To determine the in vivo persistency of the anti-NY-ESO-1 TCR-transduced T cells.

ELIGIBILITY:
* Inclusion Criteria:

  1. Must be pathology or cytology confirmed cancer patients with age of one year old and over；
  2. Must be HLA-A2 positive, and cancer tissues express NY-ESO-1；
  3. There is at least one measurable disease: diameter ≥20mm or spiral CT≥10mm；
  4. Willing to sign a durable power of attorney；
  5. Able to understand and sign the Informed Consent Document；
  6. Performance status：ECOG 0-2；
  7. Life expectancy：More than 3 months；
  8. Patients must be willing to practice birth control for four months after receiving a lymphodepleting preconditioning regimen；
  9. Patients with no pregnancy and lactation；
  10. Hematopoietic： (1) Absolute neutrophil count > 1000/mm3 without support of filgrastim； (2) Platelet count > 100,000/mm3； (3) Hemoglobin > 8.0 g/dL； (4) lymphocyte count >500/mm3； (5) WBC > 3,000/mm3；
  11. Chemistry： (1) AST and ALT < 2.5 times upper limit of normal； (2) Serum creatinine≤1.6 mg/dl； (3) Bilirubin ≤1.5 mg/dL（3.0 mg/dL in patients with Gilbert's syndrome）；
  12. Seronegative for hepatitis B and C viruses；
  13. Seronegative for human immunodeficiency virus (HIV) antibody；
  14. More than four weeks must have elapsed since any prior systemic therapy at the time of randomization, and patients' toxicities must have recovered to a grade 1 or less (except for alopecia or vitiligo). Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria；
  15. Six weeks must have elapsed since any prior anti-CTLA4 antibody therapy to allow antibody levels to decline. Patients who have previously received any anti-CTLA4 antibody and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.
* Exclusion Criteria:

  1. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease)；
  2. Active systemic infections；
  3. Coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system；
  4. Concurrent use of systemic steroids；
  5. History of severe immediate hypersensitivity reaction to any of the agents used in this study；
  6. There are obvious dysfunctions in heart , liver，kidney and other vital organs
  7. T cell lymphoma and leukemia patients；
  8. HIV positive；
  9. History of coronary revascularization or ischemic symptoms；
  10. Documented Left Ventricular Ejection Fraction (LVEF) of less than or equal to 45 percent tested in patients with: Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block；
  11. Documented forced expiratory volume 1 (FEV1) less than or equal to 60 percent predicted tested in patients with a prolonged history of cigarette smoking (20 pk/yrs of smoking) or symptoms of respiratory dysfunction；
  12. Bronchial lesions (probably shifted obstructive pneumonia or intracranial hemorrhage risk)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 8 weeks
  To evaluate the safety and feasibility of the administration of anti-NY-ESO-1 TCR transduced T cells in patients with HLA-A2+ NY-ESO-1-expressing malignancies.

SECONDARY OUTCOMES:
Number of participants with Clinical responses | 2 years
  To determine if the treatment can result in clinical regression of malignant tumors in the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, The First Affiliated Hospital of Shenzhen University, Shenzhen, Guangdong, China